CLINICAL TRIAL: NCT01848613
Title: Randomized Cross-over Study of Patient Preference for Oral or Intravenous Vinorelbine in the Treatment of Advanced NSCLC. A Phase IV Study.
Brief Title: Study of Patient Preference for Oral or Intravenous Vinorelbine in the Treatment of Advanced NSCLC
Acronym: VIVOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST162.05; 2012-003544-68 (EudraCT Number)
Record Dates: First submitted 2013-04-26; First posted 2013-05-07 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): •Arm A: first cycle of IV vinorelbine (30 mg/m2) and second cycle of PO vinorelbine (60mg/m2)
  Interventions: Drug: Vinorelbine
- Arm B (Experimental): • Arm B: first cycle with PO vinorelbine (60mg/m2) followed by a second cycle of IV vinorelbine (30mg/m2)
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine

SUMMARY:
Title: Randomized cross-over study of patient preference for oral or intravenous vinorelbine in the treatment of advanced NSCLC. A phase IV study.

ShortTitle/ Acronym: VIVOS

Protocol Code :IRST162.05

Study Design: Randomized, open label cross-over study

Study Duration: Two years

Study Center(s): Multicenter study

Objectives:

Primary: Patient preference for oral or intravenous vinorelbine Secondary: Overall Response Rate, Time to Progression, Toxicity, Survival, Subjective reasons for treatment choice.

Number of Subjects: 120

Diagnosis and Main Inclusion Criteria:

Patients affected by stage IIIB or stage IV NSCLC candidates to receive a first line chemotherapy with vinorelbine due to age ≥ 70 and Eastern Cooperative Oncology Group (ECOG) Performance status ≤2 or age ≤ 70 but ECOG PS ≥ 2

Study Product, Dose, Route, Regimen and duration of administration :

* Arm A: first cycle of IV vinorelbine (30 mg/m2) and second cycle of PO vinorelbine (60mg/m2)
* Arm B: first cycle with PO vinorelbine (60mg/m2) followed by a second cycle of IV vinorelbine (30mg/m2) In both arms vinorelbine will be given at day 1 and day 8 every 3 weeks. From the third cycle onwards patients will have to choose to receive oral or intravenous vinorelbine. Vinorelbine capsules will be administered at the dosage of 60 mg/m2 for the first course and then may be increased to 80 mg/m² at physician's choice.

Treatment will be repeated every 21 days and continued until disease progression, intolerable toxicity or patient refusal.

Reference therapy: Vinorelbine 30 mg/m2 intravenous day 1 and 8 every 21 days

Statistical Methodology: The sample size is calculated based on 75% of patients preferring "oral" vinorelbine and 25% preferring "intravenous" vinorelbine. Therefore, the investigators would compare patients preferring "oral" vinorelbine as 75% compared to a null hypothesis of 50% (no difference in proportion of patients preferring "oral" to "intravenous"). With 80% power and a total alpha of 0.05, the estimated sample size is 60 for group (120 total). During recruitment period, a formal interim analysis was planned when 60 patients (30 for group) have been enrolled, with a p-value <0.0001. To claim statistical significance in the final analysis, the overall p-value is still 5% (referred to Peto-Haybittle rule).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IIIB or IV NSCLC.
2. Age ≥ 70 and Eastern Cooperative Oncology Group (ECOG) Performance status ≤2 or age ≤ 70 but ECOG PS ≥ 2
3. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See section 9.2 and Appendix E for the evaluation of measurable disease.
4. Patients with asymptomatic brain metastases are eligible
5. Patients with recurrent disease after previous surgery are eligible
6. Life expectancy > 3 months
7. Patients must have normal organ and marrow function
8. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
9. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

1. Patients who have had previous chemotherapy for lung cancer or radiotherapy on target lesions.
2. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
3. Presence of infection.
4. Preexisting clinically significant peripheral neuropathy.
5. History or evidence of malabsorption syndrome or disease that may significantly affect gastrointestinal function.
6. Patients with known symptomatic uncontrolled brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to vinorelbine or other agents used in the study.
8. Presence of medical problems of sufficient severity to prevent full compliance with the study.
9. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Patients preference for IV or PO vinorelbine. | 2 years
  At the time of patient preference, a questionnaire will be filled in by patients.

SECONDARY OUTCOMES:
Overall response rate (RR) | 2 years
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Toxicity of both drug formulations | 2 years
Subjective reasons for treatment choice | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Dazzi, MD, Study Chair — UO Oncologia Medica, Ospedale S.Maria delle Croci, RAVENNA - ITALY
Locations (8):
- Italy (8):
  - Irccs Irst, Meldola (FC), FC
  - U.O. Oncologia Ospedale Civile degli Infermi, Faenza, RA
  - U.O. Oncologia Ospedale Civile Umberto I, Lugo, RA
  - UO Oncologia Medica, Ospedale S.Maria delle Croci, Ravenna, RA
  - U.O. Oncologia Ospedale Cervesi, Cattolica, RN
  - U.O. Oncologia ed Ematologia Oncologica ULSS 13 MIRANO, Mirano, VE
  - U.O. Oncologia Medica ULSS 1 Belluno, Belluno
  - U.O. Oncologia Ospedale degli Infermi, Rimini